CLINICAL TRIAL: NCT00659646
Title: A Randomized, Controlled, Open Label Study of the Safety and Efficacy of a Topical Gentamicin Collagen Sponge Combined With An Antibiotic Compared to Antibiotic Therapy Alone in Diabetic Patients With Moderately Infected Foot Ulcers
Brief Title: The Safety and Efficacy of an Antibiotic Sponge in Diabetic Patients With Moderately Infected Foot Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innocoll (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INN-TOP-003
Record Dates: First submitted 2008-04-11; First posted 2008-04-16 (Estimated); Results first posted 2021-08-30 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes; ulcers; ulcerations; infection
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Ulcer; Infections | interventions — Levofloxacin; Ofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Gentamicin sponge applied into wound plus levofloxacin, 750 mg by mouth (po) or intravenous (IV) every 24 hours or, if ulcer culture results show resistance to levofloxacin, alternative antimicrobial therapy as determined by susceptibility testing
  Interventions: Drug: gentamicin-collagen sponge and levofloxacin
- B (Active Comparator): Levofloxacin, 750 mg po or IV every 24 hours or, if ulcer culture results show resistance to levofloxacin, alternative antimicrobial therapy as determined by susceptibility testing
  Interventions: Drug: Levofloxacin only

INTERVENTIONS:
Drug: gentamicin-collagen sponge and levofloxacin — Topical Gentamicin Collagen Sponge: 10 × 10 cm in size And 750 mg tablet po every 24 hours or 750 mg IV administered by slow infusion over 90 minutes every 24 hours.
  Other Names: Collatamp G
  Arms: A
Drug: Levofloxacin only — levofloxacin, 750 mg tablet po every 24 hours or 750 mg IV administered by slow infusion over 90 minutes every 24 hours
  Other Names: Tavanic, Levaquin
  Arms: B

SUMMARY:
The purpose of this study is to determine whether the gentamicin-collagen sponge when combined with standard daily wound care and an oral antibiotic (levofloxacin) is safe and effective in treating moderately infected skin ulcers compared to treatment only with standard daily wound care and an oral antibiotic (levofloxacin).

DETAILED DESCRIPTION:
Infected skin ulcers with diabetes can be very debilitating because they are difficult to heal. Diabetic ulcers are responsible for frequent health care visits, and are a major predictor of amputation. Diabetic ulcers can be caused by a patient's inability to sense pain or warmth as well as peripheral vascular disease, which causes diminished blood flow to the foot. Early aggressive treatment is necessary to treat infection and ultimately prevent the need for amputation.

Gentamicin is an antibiotic that is effective in treating certain kinds of infection. Collagen is a protein that is found in all mammals. The gentamicin-collagen sponge is a thin flat sponge made out of collagen that comes from cow tendons and containing gentamicin. When applied to an open ulcer, the collagen breaks down and the gentamicin is released into the ulcer, but very little is absorbed into the blood stream. The high levels of gentamicin in the open infected ulcer may help treat the infection.

In this study, all subjects will be given the necessary supplies and taught how to take care their foot ulcer. All subjects will also receive oral an antibiotic (levofloxacin). Additionally, subjects who are randomly assigned to receive the gentamicin-collagen sponge will place a gentamicin-collagen sponge on their ulcer during daily wound care.

ELIGIBILITY:
Inclusion Criteria:

* Is a man or woman aged ≥ 18 and ≤ 80 years.
* Has diabetes mellitus, according to the American Diabetes Association criteria.
* Has a single infected skin ulcer below the knee, defined as "moderate" by the Infectious Disease Society of America (IDSA) Guidelines for whom, in the Investigator's opinion, intravenous (IV) or oral antimicrobial therapy is appropriate
* Has had an x ray of the infected area within the 2 days immediately preceding or at Visit 1 (Baseline/Randomization) to document the presence or absence of osteomyelitis. Patients with osteomyelitis must receive appropriate surgical intervention to remove all necrotic and infected bone and otherwise meet enrollment criteria before being enrolled in the study.
* Meets certain minimal laboratory criteria
* Has an ankle brachial index (ABI) > or = 0.7 and ≤ 1.3. (Note: Patients with ABI < 0.7 or > 1.3 may be included if they have either a transcutaneous oxygen pressure or a toe pressure > or = 40 mm Hg on limb with ulcer.)
* If female, is nonpregnant (negative pregnancy test results at the Baseline/Randomization Visit) and nonlactating.
* If female, is either not of childbearing potential (defined as postmenopausal for ≥ 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy or hysterectomy]) or practicing a medically acceptable methods of birth control and agrees to continue with the regimen throughout the study
* Willing to return to the study facility for the Final Study Visit.
* Must be able to fluently speak and understand English and be able to provide meaningful written informed consent for the study.

Exclusion Criteria:

* Has a known history of hypersensitivity to gentamicin (or other systemic aminoglycosides) or levofloxacin or drugs in the same class, or any of the test article or reference product components.
* Has a known hypersensitivity to bovine collagen.
* Has any uncontrolled illnesses that, in the opinion of the Investigator, would interfere with interpreting the results of the study.
* Has a target ulcer with a wound size > 10 × 10 cm.
* Has gangrenous tissue of the affected limb that cannot be removed with a single debridement.
* Has wound known to contain isolates resistant to levofloxacin.
* Has a wound associated with prosthetic material or device.
* Received any topical or systemic antimicrobial therapy within the 2 weeks prior to study entry (Visit 1 [Day 1]).
* If severely immunocompromised, may be excluded at the discretion of the Investigator.
* Has a history of alcohol or substance abuse in the past 12 months.
* Has serum creatinine > 3 mg/dL, is undergoing dialysis (renal or peritoneal) or has a history of kidney transplant.
* Has a history of myasthenia gravis or other neurological condition where gentamicin use is contraindicated as determined by the Investigator.
* Has a history of epilepsy
* Has a history of tendon disorders related to fluoroquinolone administration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Prior, Study Director — Innocoll
Locations (1):
- Karr Foot Kare PA, Lakeland, Florida, United States

REFERENCES:
- [Result] Lipsky BA, Kuss M, Edmonds M, Reyzelman A, Sigal F. Topical application of a gentamicin-collagen sponge combined with systemic antibiotic therapy for the treatment of diabetic foot infections of moderate severity: a randomized, controlled, multicenter clinical trial. J Am Podiatr Med Assoc. 2012 May-Jun;102(3):223-32. doi: 10.7547/1020223. PMID 22659765

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Investigative medical sites
Groups:
- Levofloxacin: Levofloxacin only: levofloxacin, 750 mg tablet po every 24 hours or 750 mg IV administered by slow infusion over 90 minutes every 24 hours
Period: Overall Study
Arm/Group | Gentamicin-collagen Sponge and Levofloxacin | Levofloxacin
Started | 38 | 18
Completed | 23 | 10
Not Completed | 15 | 8
Not completed — Protocol Violation | 12 | 8
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — protocol noncompliance after randomized | 1 | 0

BASELINE CHARACTERISTICS:
Population: modified intent-to-treat
Groups:
- Gentamicin Sponge: Gentamicin sponge applied into wound plus levofloxacin, 750 mg by mouth (po) or intravenous (IV) every 24 hours or, if ulcer culture results show resistance to levofloxacin, alternative antimicrobial therapy as determined by susceptibility testing
  gentamicin-collagen sponge and levofloxacin: Topical Gentamicin Collagen Sponge: 10 × 10 cm in size And 750 mg tablet po every 24 hours or 750 mg IV administered by slow infusion over 90 minutes every 24 hours.
- Levofloxacin: Levofloxacin, 750 mg po or IV every 24 hours or, if ulcer culture results show resistance to levofloxacin, alternative antimicrobial therapy as determined by susceptibility testing
  Levofloxacin only: levofloxacin, 750 mg tablet po every 24 hours or 750 mg IV administered by slow infusion over 90 minutes every 24 hours
- Total: Total of all reporting groups
Arm/Group | Gentamicin Sponge | Levofloxacin | Total
Number analyzed (Participants) | 26 | 10 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (9.17) | 55.1 (14.3) | 59.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 11
  Male | 17 | 8 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 10 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Clinical Cure at Visit 3 (Day 7)
Description: Number of participants with a clinical cure in each treatment group at Visit 3 (Day 7). Clinical Cure is defined as positive clinical response and with pathogen eradication.
Time Frame: Day 7 of treatment
Population: modified intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Sponge | Levofloxacin
Number analyzed (Participants) | 26 | 10
Participants | 0 | 3

2. Secondary Outcome: Number of Participants With a Positive Clinical Response at Each Time Point
Description: Number of patients with positive clinical response, defined as those with a clinical outcome of "clinical cure" or "clinical improvement" in each treatment group at/by each time point
Time Frame: Day 3, 7, 10,14, 21, 28 and 42
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Sponge | Levofloxacin
Number analyzed (Participants) | 26 | 10
Participants
  Visit 2 Day 3 | 24 | 9
  Visit 3 Day 7 | 26 | 10
  Visit 4 Day 10 | 25 | 7
  Visit 5 Day 14 | 24 | 6
  Visit 6 Day 21 | 14 | 3
  Visit 7 Day 28 | 10 | 3
  Final Study Visit Day 42 | 22 | 10

3. Secondary Outcome: Number of Participants With a Clinical Cure at Each Visit Except Visit 3 (Day 7)
Description: clinical cure is defined as having a positive clinical response and with pathogen eradication
Time Frame: Day 3, 10, 14, 21, 28 & 42
Population: mITT
Measure: Count of Participants; unit: Participants
Groups:
- No Sponge: Levofloxacin, 750 mg po or IV every 24 hours or, if ulcer culture results show resistance to levofloxacin, alternative antimicrobial therapy as determined by susceptibility testing
  Levofloxacin only: levofloxacin, 750 mg tablet po every 24 hours or 750 mg IV administered by slow infusion over 90 minutes every 24 hours
Arm/Group | Gentamicin Sponge | No Sponge
Number analyzed (Participants) | 26 | 10
Participants
  Visit 2 Day 3 | 0 | 0
  Visit 4 Day 10 | 1 | 0
  Visit 5 Day 14 | 10 | 3
  Visit 6 Day 21 | 4 | 0
  Visit 7 Day 28 | 9 | 1
  Final Visit Day 42 | 22 | 7

4. Secondary Outcome: Number of Participants With Pathogen Eradication by Visit
Time Frame: Day 3, 7, 10, 14, 21 & 28
Population: mITT
Measure: Count of Participants; unit: Participants
Groups:
- No Sponge: No Sponge
  Levofloxacin, 750 mg po or IV every 24 hours or, if ulcer culture results show resistance to levofloxacin, alternative antimicrobial therapy as determined by susceptibility testing
  Levofloxacin only: levofloxacin, 750 mg tablet po every 24 hours or 750 mg IV administered by slow infusion over 90 minutes every 24 hours
Arm/Group | Gentamicin Sponge | No Sponge
Number analyzed (Participants) | 26 | 8
Participants
  Visit 2 Day 3 | 20 | 1
  Visit 3 Day 7 | 24 | 2
  Visit 4 Day 10 | 23 | 2
  Visit 5 Day 14 | 18 | 2
  Visit 6 Day 21 | 12 | 0
  Visit 7 Day 28 | 5 | 0

5. Secondary Outcome: Change From Baseline in Total Wound Surface Area Measured in cm^2
Description: Wound Surface Area was measured in cm² Actual Values Total wound surface area was compared across treatments using 2-sample t-tests. Wound tracings were obtained at study visits by trained study personnel who were blinded to the patient data and regimen. A centralized imaging facility provided both wound perimeter and area measurements.
Time Frame: Day 3, 7, 10, 14, 21, 28 & 42
Population: mITT
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Gentamicin Sponge | No Sponge
Number analyzed (Participants) | 26 | 10
cm^2
  Visit 1 Day 1 | 5.11 (9.249) | 1.24 (0.998)
  Visit 2 Day 3 | 4.50 (8.53) | .92 (.78)
  Visit 3 Day 7 | 4.47 (8.19) | .76 (.707)
  Visit 4 Day 10 | 4.31 (8.730) | 1.14 (0.760)
  Visit 5 Day 14 | 4.14 (9.041) | 0.95 (.656)
  Visit 6 Day 21 | 2.93 (5.517) | 1 (0.671)
  Visit 7 Day 28 | 2.67 (5.474) | .93 (0.606)
  Final Study Visit Day 42 | 3.73 (9.047) | .64 (.846)

6. Secondary Outcome: Time to Clinical Cure
Description: clinical cure is defined as having a positive clinical response and with pathogen eradication
Time Frame: Days 1 through 49
Population: mITT
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Gentamicin Sponge | No Sponge
Number analyzed (Participants) | 26 | 10
Days | 21 [14.0 to 28.0] | 14 [7.0 to 40.0]

7. Secondary Outcome: Visual Analog Scale (VAS) for Pain Assessment
Description: Measured on a Visual Analog Pain Scale (VAS) with the lowest possible value of 0 and highest 100 (0 - 100) at each time point. A lower score is better which means the patient experience lower pain. The score is calculated using the number of hours * the VAS score. This represents the AUC (Area Under the Curve) of the pain intensities when calculated with the trapezoidal rule. For each measure outcome - the minimum score is "0" and the maximum score is 100* the number of hours in that period.
Time Frame: Day 3, 7, 10, 14, 21, 28 & 42
Measure: Mean (Standard Deviation); unit: score on a scale*days
Arm/Group | Gentamicin Sponge | No Sponge
Number analyzed (Participants) | 26 | 10
score on a scale*days
  Visit 1 Day 1 | 39.2 (36.79) | 26.3 (21.77)
  Visit 2 Day 3 | 27.6 (32.22) | 18.7 (19.60)
  Visit 3 Day 7 | 17.5 (23.58) | 12.6 (19.67)
  Visit 4 Day 10 | 17.2 (23.34) | 13.6 (20.98)
  Visit 5 Day 14 | 13.3 (20.99) | 13.2 (21.45)
  Visit 6 Day 21 | 22.9 (34.20) | 14.3 (22.28)
  Visit 7 Day 28 | 14.3 (30.96) | 9.3 (10.07)
  Final Study Visit Day42 | 17.3 (28.84) | 2.3 (28.84)

8. Secondary Outcome: Lipsky Wound Score
Description: The Lipsky wound scoring scale consists of scoring categories for purulent drainage, non-purulent drainage, erythema, induration, tenderness, pain, local warmth and wound measurements. This wound scoring system allows us to take the size and depth of the wound into consideration as well as all signs and symptoms of inflammation and infection. A quantitative score that assess wounds both at baseline and during therapy to compare wound scores over time. The higher the score the worse the inflammation and/or infection is. The Lowest score possible is "3" and the highest score possible is "64".
Time Frame: Days 3, 7, 10, 14, 21, 28, 42
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gentamicin Sponge | No Sponge
Number analyzed (Participants) | 24 | 10
score on a scale
  Visit 1 Day 1 | 17.67 (4.498) | 13.10 (5.043)
  Visit 2 Day 3 | 13.58 (4.373) | 11 (3.771)
  Visit 3 Day 7 | 10.79 (4.364) | 7.60 (4.300)
  Visit 4 Day 10 | 9.17 (4.108) | 8.29 (3.147)
  Visit 5 Day 14 | 8.36 (4.315) | 5.33 (1.633)
  Visit 6 Day 21 | 7.29 (3.970) | 4.33 (2.309)
  Visit 7 Day 28 | 5.10 (2.87) | 3.67 (1.155)
  Final Study Visit Day 42 | 6.18 (4.239) | 4.80 (2.251)

ADVERSE EVENTS:
Time Frame: Day 42
Arm/Group | Gentamicin Sponge | Levofloxacin
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/18
Serious Adverse Events (participants affected / at risk) | 5/38 | 1/18
Other Adverse Events (participants affected / at risk) | 4/38 | 1/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gentamicin Sponge (N=38) | Levofloxacin (N=18)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Wound haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gentamicin Sponge (N=38) | Levofloxacin (N=18)
Tinea pedis (Infections and infestations) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other